CLINICAL TRIAL: NCT05776238
Title: Lateral Position for Premature Babies Undergone Sedation During Magnetic Resonance Imaging: an Observational Study
Brief Title: Lateral Position MRI in Preterm Infants, an Observational Study
Acronym: MRIOPS
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5259B
Record Dates: First submitted 2023-02-17; First posted 2023-03-20 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-02

CONDITIONS: Prematurity; Magnetic Field Exposure; Sedation Complication
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate safety of sedation in lateral position in premature babies undergone MRI. The main question it aims to answer are:

* number of apneas during sedation
* Maintenance of eupnea during deep sedation

DETAILED DESCRIPTION:
Premature babies will be sedated in lateral position during Magnetic Resonance Imaging. During procedure we provide a close control about eupnea maintenance (SaO2 and EtCO2) in order to verify the safety of laying.

ELIGIBILITY:
Inclusion Criteria:

* < 40 weeks Post Conceptional Age (PCA)

Exclusion Criteria:

* > 50 weeks PCA
* previous treatment with hypothermia for neonatal asphyxia
* patients who received invasive positive pressure ventilation within the previous 48 h
* preexisting cardiac arrhythmias
* presence or suspicion of oncological pathology
* neuromuscular or metabolic diseases
* previous brain or abdominal surgery
* presence of epicranial venous accesses
* upper respiratory tract infections
* refusal of informed consent by parents or inability to express it

Max Age: 50 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Prematures babies during in hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Peripheral oxygen desaturation | Through study completion, an average of 7 month
  Number of episodes of peripheral oxygen desaturation < 90% during deep sedation
Apnea | Through study completion, an average of 7 month
  Number of episodes of apnea > 20 sec during deep sedation

SECONDARY OUTCOMES:
Subjective evaluation of imaging quality | Through study completion, an average of 7 month
  Subjective evaluation of images by two neuroradiologists measured as Score (1-5 points) in 5 categories
Objective evaluation of imaging quality | Through study completion, an average of 7 month
  Objective evaluation of image quality by measuring the Signal to Noise Ratio (SNR)
Post-operative temperature control | Through study completion, an average of 7 month
  Measurement of rectal core body temperature (°C) after the exam
Time for full enteral feeding | Through study completion, an average of 7 month
  How many hours for full enteral feeding after the preoperative fasting
Objective evaluation of imaging quality | Through study completion, an average of 7 month
  Objective evaluation of image quality by measuring the Contrast to Noise Ratio (CNR)

CONTACTS AND LOCATIONS:
Overall Officials: fabio sbaraglia, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Policlinico Univeristario Agostino Gemelli, Roma, Rome, Italy

REFERENCES:
- [Derived] Sbaraglia F, Gaudino S, Tiberi E, Maiellare F, Spinazzola G, Garra R, Della Sala F, Micci DM, Russo R, Riitano F, Ferrara G, Vento G, Rossi M. Deep sedation in lateral position for preterm infants during cerebral magnetic resonance imaging: a pilot study. J Anesth Analg Crit Care. 2024 Dec 18;4(1):80. doi: 10.1186/s44158-024-00216-9. PMID 39696670